CLINICAL TRIAL: NCT05603559
Title: Safety, Dosimetry and Dose-escalation of 177Lu-P17-087/177Lu-P17-088 in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: 177Lu-P17-087/177Lu-P17-088 in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUMCH-NM-087/088
Record Dates: First submitted 2022-10-25; First posted 2022-11-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 177Lu-P17-087 arm (Experimental): All patients were intravenous injected with single dose 1.1 GBq (30 mCi) of 177Lu-P17-087 then monitored at 1.5 hours, 4 hours, 24 hours, 48 hours, 72 hours, 120 hours and 168 hours post-injection.
  Interventions: Drug: 1.1 GBq (30 mCi) of 177Lu-P17-087
- 177Lu-P17-088 arm (Experimental): All patients were intravenous injected with single dose 1.1 GBq (30 mCi) of 177Lu-P17-088 then monitored at 1.5 hours, 4 hours, 24 hours, 48 hours, 72 hours, 120 hours and 168 hours post-injection.
  Interventions: Drug: 1.1 GBq (30 mCi) of 177Lu-P17-088

INTERVENTIONS:
Drug: 1.1 GBq (30 mCi) of 177Lu-P17-087 — All patients were intravenous injected with single dose 1.1 GBq (30 mCi) of 177Lu-P17-087 then monitored at 1.5 hours, 4 hours, 24 hours, 48 hours, 72 hours, 120 hours and 168 hours post-injection.
  Arms: 177Lu-P17-087 arm
Drug: 1.1 GBq (30 mCi) of 177Lu-P17-088 — All patients were intravenous injected with single dose 1.1 GBq (30 mCi) of 177Lu-P17-088 then monitored at 1.5 hours, 4 hours, 24 hours, 48 hours, 72 hours, 120 hours and 168 hours post-injection.
  Arms: 177Lu-P17-088 arm

SUMMARY:
This is a pilot study to assess the safety and measure image-based absorbed dose of 177Lu-P17-087/177Lu-P17-088 in patients with metastatic castration-resistant prostate cancer (mCRPC) who will undergo radioliagnd therapy using 177Lu-P17-087/177Lu-P17-088. All patients underwent whole-body 68Ga-PSMA PET/CT for selection and accepted intravenous injection with single dose 1.1 GBq (30 mCi) of 177Lu-P17-087/177Lu-P17-088 within one week, then monitored at 1.5 hours, 4 hours, 24 hours, 48 hours, 72 hours, 120 hours and 168 hours after 177Lu-P17-087/177Lu-P17-088 administration with serial whole body planar and SPECT/CT imaging.Following this initial safety assessment, the study will proceed to a dose-escalation phase designed to further evaluate safety and determine the optimal therapeutic activity. The dose-escalation phase will enroll patients into three sequential cohorts: a 1.11 GBq (30 mCi) dose group, a 2.96 GBq (80 mCi) dose group, and a 4.44 GBq (120 mCi) dose group.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent malignant tumor in men worldwide. Prostate-specific membrane antigen (PSMA), is a surface molecule specifically expressed by prostate tumors which was shown to be a valid target for radiotherapy. 177Lu-PSMA-617, a urea-based compound, provide an effective target for the treatment of metastatic castration-resistant prostate cancer. However, a major problem in the therapeutic use of 177Lu-PSMA-617 has been its short half-life and fast rate of clearance. The investigators designed and synthesized a new radiopharmaceutical based on PSMA-11, P16-093. 68Ga-P16-093 showed higher tumor uptake and clear blood clearance than 68Ga-PSMA-617. Then, the investigators shynthesis a new therapeutic radiopharmaceutical based on P16-093, P17-087; and the investigators added a selected albumin binder into P17-088 to synthesis another new radiopharmaceutical, P17-088. This study is designed to evaluate the safety, dosimetry, and preliminary antitumor activity of 177Lu-P17-087/177Lu-P17-088. The trial will include an initial dose-escalation phase to identify the maximum tolerated dose (MTD) or optimal biological dose, which will be followed by a dose-expansion phase to confirm safety and further characterize pharmacokinetics and efficacy, thereby establishing the Recommended Phase II Dose (RP2D) for future development.

ELIGIBILITY:
Inclusion Criteria:

* All the patients had progressive metastatic castration-resistant prostate cancer that did not respond to androgen-suppression therapy and/or systemic chemotherapy;
* Distant metastases with high PSMA expression were confirmed on 68Ga-PSMA PET/CT within one week before the injection of 177Lu-P17-087/177Lu-P17-088.

Exclusion Criteria:

* Patients were excluded if they had [18F]FDG positive tumors without corresponding PSMA uptake. Patients were also not eligible if they accepted other radionuclide therapies within 6 months or had clinically significant impaired bone marrow, liver, or kidney function with a hemoglobin level of less than 9.0 g/dL, a white blood cell count of less than 2.5×109/L, a platelet count of less than 100×109/L and a serum creatinine > 100 μmol/L.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
Dosimetry of normal organs and tumors | Determined using imaging at 1.5 hours, 4 hours, 24 hours, 48 hours, 72 hours, 120 hours and 168 hours after the first administration of 177Lu-P17-087/088
  The semiquantitative dosimetry will be performed based on SPECT/CT acquisitions after the administration of 177Lu-P17-087/177Lu-P17-088. The dose delivered to normal organs and tumors will be recorded.
Hematologic adverse events collection | through study completion, an average of 2 weeks
  Hematologic status were performed before and every 2 weeks after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.
Hepatic and renal toxic events collection | through study completion, an average of 2 weeks
  Liver function, and renal function were performed before and 6 weeks after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
PSA Response | through study completion, an average of 3 weeks
  The serum PSA response was documented semimonthly until 6 weeks after the administration of 177Lu-P17-087/177Lu-P17-088. PSA response was classified as the following: partial response (PR) if PSA decrease ≥50%, progressive disease (PD) if PSA increase ≥ 25% and stable disease (SD) if PSA increase <25% or PSA decrease <50%.
PSMA Response | 6 weeks after treatment administration.
  Treatment efficacy will be assessed by comparing PSMA-expression on PET/CT at baseline to the scan obtained at the 6-week follow-up. Tumor response will be evaluated according to the RECIP 1.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li L, Wang J, Wang G, Wang R, Jin W, Zang J, Sui H, Jia C, Jiang Y, Hong H, Zhu L, Alexoff D, Ploessl K, Kung HF, Zhu Z. Comparison of novel PSMA-targeting [177Lu]Lu-P17-087 with its albumin binding derivative [177Lu]Lu-P17-088 in metastatic castration-resistant prostate cancer patients: a first-in-human study. Eur J Nucl Med Mol Imaging. 2024 Jul;51(9):2794-2805. doi: 10.1007/s00259-024-06721-x. Epub 2024 Apr 25. PMID 38658392